CLINICAL TRIAL: NCT05252364
Title: A Phase 1 Open-Label Study to Assess the Safety, Pharmacokinetics, and Anti-tumor Activity of Oral HP518 in Patients With Metastatic Castration-Resistant Prostate Cancer
Brief Title: A Study to Assess the Safety, Pharmacokinetics, and Anti-Tumor Activity of Oral HP518 in Patients With Metastatic Castration-Resistant Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hinova Pharmaceuticals Aus Pty Ltd (Industry)
Responsible Party: Sponsor
Organization: Hinova Pharmaceuticals Inc. (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HP518-CS-001
Record Dates: First submitted 2021-12-03; First posted 2022-02-23 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Metastatic Castration-resistant Prostate Cancer

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Part 1 - Dose Escalation, 25mg/d (Cohort 1) (Experimental): Oral tablet(s), once daily in 28-day cycles
  Interventions: Drug: HP518 - Dose Escalation
- Part 1 - Dose Escalation 100mg/d (Cohort 2) (Experimental): Oral tablet(s), once daily in 28-day cycles
  Interventions: Drug: HP518 - Dose Escalation
- Part 1 - Dose Escalation 200mg/d (Cohort 3) (Experimental): Oral tablet(s), once daily in 28-day cycles
  Interventions: Drug: HP518 - Dose Escalation
- Part 1 - Dose Escalation 300mg/d (Cohort 4) (Experimental): Oral tablet(s), once daily in 28-day cycles
  Interventions: Drug: HP518 - Dose Escalation
- Part 1 - Dose Escalation 400mg/d (Cohort 5) (Experimental): Oral tablet(s), once daily in 28-day cycles
  Interventions: Drug: HP518 - Dose Escalation
- Part 1 - Dose Escalation 500mg/d (Cohort 6) (Experimental): Oral tablet(s), once daily in 28-day cycles
  Interventions: Drug: HP518 - Dose Escalation
- Part 2 - Dose Expansion (Experimental): Oral tablet(s), once daily in 28-day cycles
  Interventions: Drug: HP518 - Dose expansion

INTERVENTIONS:
Drug: HP518 - Dose Escalation — Part 1: Dose escalation
  Daily oral dosage with the prescribed dose level based on Cohort assignment.
  Arms: Part 1 - Dose Escalation 100mg/d (Cohort 2); Part 1 - Dose Escalation 200mg/d (Cohort 3); Part 1 - Dose Escalation 300mg/d (Cohort 4); Part 1 - Dose Escalation 400mg/d (Cohort 5); Part 1 - Dose Escalation 500mg/d (Cohort 6); Part 1 - Dose Escalation, 25mg/d (Cohort 1)
Drug: HP518 - Dose expansion — Part 2: Dose expansion
  Daily oral dosage with the highest dose with acceptable toxicity (RP2D) based on data from Part 1.
  Arms: Part 2 - Dose Expansion

SUMMARY:
The overall objective of this Phase 1 study is to evaluate the safety, PK, and anti-tumor activity of 12 weeks of daily oral dosing with HP518 after selecting the RP2D of HP518 based on assessments of multiple dose escalation in patients with progressive mCRPC.

DETAILED DESCRIPTION:
This First in Human dose escalation and expansion study of HP518 in patients with mCRPC is being conducted not only to evaluate the safety and tolerability of orally administered HP518, but also to provide necessary information for efficacy analysis in future studies.

ELIGIBILITY:
Inclusion Criteria:

1. Has histologically confirmed adenocarcinoma of the prostate.
2. Has metastatic disease at study entry documented by 2 or more bone lesions on bone scan or by soft tissue disease observed by CT/MRI.
3. Has disease progression while receiving any ADT, androgen biosynthesis inhibitors, or second-generation AR inhibitors.
4. Must have recovered from toxicities related to any prior treatments
5. Ongoing ADT with LHRH agonist/antagonist therapy or history of bilateral orchiectomy.
6. ECOG performance status score of 0 to 1.

Exclusion Criteria:

1. Has received more than 1 line of chemotherapy for prostate cancer.
2. Use of enzalutamide, and/or other second-generation AR inhibitors and/or abiraterone as follows:

   * Received any agent within 4 weeks prior to the start of study drug.
   * Discontinued agent without evidence of radiographic or PSA progression.
3. Has had any anticancer treatments, including immunotherapy, chemotherapy, or radiotherapy (eg, 177Lu-PSMA-617, radium 223, PARP inhibitor) within 4 weeks prior to the first dose of HP518.
4. Has gastrointestinal disorder affecting absorption (e.g., gastrectomy).
5. Has significant cardiovascular disease.
6. Use of an investigational agent, without evidence of radiographic or PSA progression, within 4 weeks prior to the first dose of HP518 or a period required by local regulation, whichever is longer.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 22 (Actual)
Dates: Start 2021-12-14 (Actual); Primary Completion 2024-01-22 (Actual); Study Completion 2024-01-22 (Actual)

PRIMARY OUTCOMES:
Incidences of Protocol-defined DLT during the DLT assessment period , characterized by type, frequency, severity (as graded by NCI CTCAE version 5.0), timing, seriousness, and relationship to study drug | 28 days
  To evaluate the safety and tolerability and determine the MTD and the RP2D of orally administered HP518 (Part 1)
Incidence of Treatment-Emergent Adverse Events characterized by type, frequency, severity (as graded by NCI CTCAE version 5.0), timing, seriousness | Through study completion, an average of 1 year
  To evaluate the safety and tolerability and determine the MTD and the RP2D of orally administered HP518 (Part 1)
Incidence of laboratory abnormalities, characterized by type, frequency, severity (as graded by NCI CTCAE version 5.0), and timing | Through study completion, an average of 1 year
  To evaluate the safety and tolerability and determine the MTD and the RP2D of orally administered HP518 (Part 1)
Incidence of vital signs abnormalities characterized by type, frequency, severity (as graded by NCI CTCAE version 5.0), and timing | Time Frame: Through study completion, an average of 1 year
  To evaluate the safety and tolerability and determine the MTD and the RP2D of orally administered HP518 (Part 1)
Incidence of ECG (PR, QRS, QT, and QTcF intervals) abnormalities characterized by type, frequency, severity (as graded by NCI CTCAE version 5.0), and timing | Through study completion, an average of 1 year
  To evaluate the safety and tolerability and determine the MTD and the RP2D of orally administered HP518 (Part 1)
Proportion of patients showing a PSA decline of ≥50% between baseline and Week 12 of dosing with HP518. | 12 weeks

SECONDARY OUTCOMES:
Assessment of pharmacokinetic parameters of HP518 : area under the concentration-time curve (AUC) | 12 weeks
Assessment of pharmacokinetic parameters of HP518: Maximum concentration (Cmax) | 12 weeks
Assessment of pharmacokinetic parameters of HP518: Time to maximum concentration (Tmax) | 12 weeks
Assessment of pharmacokinetic parameters of HP518: apparent terminal elimination half-life (T1/2) | 12 weeks
Assessment of pharmacokinetic parameters of HP518: apparent volume of distribution during the terminal phase after extravascular administration (Vz/F) | 12 weeks
Assessment of pharmacokinetic parameters of HP518: oral clearance (CL/F) | 12 weeks
Assessment of PSA50 from baseline to after 4 and 8 weeks of dosing with HP518 | 8 weeks
  To evaluate PSA50 from baseline to after 4 and 8 weeks of dosing with HP518
Time to PSA progression using the PCWG3 definition (PSA >25% and >2 ng/mL above nadir, confirmed by progression at 2 time points at least 3 weeks apart) | Through study completion, an average of 1 year
  To evaluate the time to PSA progression
Time to radiographic progression using the RECIST v1.1 and PCWG3 definition | Through study completion, an average of 1 year
  To evaluate radiographic progression per RECIST v1.1 and PCWG3
Radiographic response measured by RECIST 1.1 in patients with measurable soft tissue disease at baseline | Through study completion, an average of 1 year
  To assess objective response by RECIST v1.1 (proportion of patients with a PR or CR) in patients with measurable soft tissue disease at baseline
Change in number of AR N-term-positive CTCs/ml from baseline to week 12 | 12 weeks
Genomic profiling using cfDNA | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Zhonghua Zhou, Study Director — Hinova Pharmaceuticals USA, Inc.
Locations (5):
- Australia (5):
  - Border Medical Oncology, Albury, New South Wales
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - Macquarie University, Macquarie Park, New South Wales
  - Peter McCallum Cancer Center, Melbourne, Victoria
  - Alfred Hospital, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Azad AA, Gurney H, Underhill C, Horvath L, Voskoboynik M, Li X, King I, Shao L, Dai Y, Perabo F. Phase 1 study of HP518, a PROTAC AR degrader in patients with mCRPC: results on safety, pharmacokinetics, and anti-tumor activity. Invest New Drugs. 2025 Apr;43(2):435-445. doi: 10.1007/s10637-025-01533-8. Epub 2025 Apr 28. PMID 40289067